CLINICAL TRIAL: NCT02871206
Title: A Randomized Controlled Trial of Adjuvanted Inactivated Vaccine Versus Inactivated Influenza Vaccine in Hutterite Children
Brief Title: Adjuvanted Inactivated Vaccine Versus Inactivated Influenza Vaccine in Hutterite Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: University of Calgary (Other); University of Saskatchewan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AV-IIV
Record Dates: First submitted 2016-08-15; First posted 2016-08-18 (Estimated); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — fluad vaccine; Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Adjuvanted Influenza Vaccine (Experimental): Fluad. A 0.25 ml intramuscular dose of the vaccine will be administered to children aged from 6 months to less than 36 months and a 0.5ml dose will be administered to children aged from 36 months to 6 years. Previously unvaccinated children who are less than 9 years of age at the time of immunization will receive a second 0.25 ml dose of the vaccine four weeks following the first vaccine as per influenza immunization recommendations if they are aged between 6 months and less than 36 months or a second dose of 0.5ml if they are aged from 36 months to 6 years.
  Interventions: Biological: Fluad
- Quadrivalent Influenza Vaccine (Active Comparator): Fluzone. A 0.5 ml dose of the vaccine will be administered intramuscularly. Previously unvaccinated children who are less than 9 years of age at the time of immunization will receive a second 0.5 ml dose of the influenza vaccine four weeks following the first vaccine as per influenza immunization recommendations.
  Interventions: Biological: Fluzone

INTERVENTIONS:
Biological: Fluad
  Arms: Adjuvanted Influenza Vaccine
Biological: Fluzone
  Arms: Quadrivalent Influenza Vaccine

SUMMARY:
This study is a randomized controlled trial (RCT) comparing adjuvanted influenza vaccine (AV) to unadjuvanted inactivated influenza vaccine (IIV). Children in Hutterite colonies in Alberta and Saskatchewan will receive AV or IIV. The goal of this study is to determine whether the AV vaccine, can provide increased community-wide protection.

ELIGIBILITY:
Group A: Receive Intervention

Inclusion Criteria:

-Healthy children aged 6 months to 72 months

Exclusion Criteria:

* Anaphylactic reaction to a previous dose of influenza vaccine or to any of its components
* Known Immunoglobulin E (IgE)-mediated hypersensitivity to eggs manifested as hives, swelling of the mouth and throat, difficulty in breathing, hypotension, or shock
* Guillain- Barré syndrome within eight weeks of a previous influenza vaccine
* Use of aspirin or salicylate- containing products within 30 days before enrollment

Group B:

Inclusion Criteria:

* household and extended family members of children in Group A
* extended family is defined as the household members of the grandparents of the children in Group A

Exclusion Criteria:

* there are no exclusion criteria for this category of participants

Group C:

Inclusion Criteria:

* other Hutterite community members that are not in Group A

Exclusion Criteria:

* there are no exclusion criteria for this category of participants

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3425 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Laboratory-confirmed influenza infection | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Mark Loeb, MD, MSc., Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Switzer C, Verschoor CP, Pullenayegum E, Singh P, Loeb M. Adjuvant-attenuated symptom severity of influenza infections in vaccinated children. Infect Med (Beijing). 2022 Sep 15;1(3):163-170. doi: 10.1016/j.imj.2022.09.002. eCollection 2022 Sep. PMID 38077624